CLINICAL TRIAL: NCT01684735
Title: Diffusion Weighted Magnetic Resonance Imaging of the Breast During Chemotherapy: Response Evaluation
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: B322201213618
Record Dates: First submitted 2012-05-14; First posted 2012-09-13 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: diffusion-weighted magnetic resonance imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women with BRCA and chemotherapy: women recently diagnosed with breast cancer and start with neo-adjuvant chemotherapy (6 cycles) before surgery/therapy

SUMMARY:
Evaluation of the response to chemotherapy in breast cancer patients by the use of Diffusion-weighted magnetic resonance imaging of the breast before the start of chemotherapy, after one and 3 cycles of therapy and at the end of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* core biopsy with diagnosis of breast cancer
* start of neo-adjuvant chemotherapy

Exclusion Criteria:

* magnetic resonance imaging incompatibility

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women diagnosed with breast cancer and treated with neo-adjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Response to chemotherapy | 1 year
  outcome is the results of pathology after chemotherapy and surgery. Data will be collected for a period of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Van Ongeval, MD, Phd, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium